CLINICAL TRIAL: NCT05459168
Title: Leveraging an Academic-Industry Partnership to Develop a Cancer-Specific Mobile Meditation App
Brief Title: Development of Calm for Cancer Prototype Mobile App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calm.com, Inc. (Industry)
Collaborators: The University of Texas Health Science Center at San Antonio (Other); Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00013029
Record Dates: First submitted 2022-03-17; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This study consists of multiple phases/aims, but within each phase/aim (excluding Aim 2 as this is just app development), there is a single group assignment. The intervention model layout described herein was the most appropriate method to describe each of the involved phases and steps.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Calm Meditation Smartphone App Feedback (Aim 1) (Other): Advisory committee members will be asked to use the current Calm meditation app platform for a full week and to keep an informal journal prior to participating in focus groups in which they will provide feedback about the app.
  Interventions: Other: Calm Meditation Smartphone App Feedback
- Cancer-Specific Meditation App Prototype Design (Aim 2) (Other): Findings from Aim 1 will inform the development of a cancer-specific meditation app prototype to be tested in Aim 3.
  Interventions: Other: Cancer-Specific Meditation App Prototype Design
- Cancer-Specific Meditation App Prototype (Aim 3) (Other): Recruited cancer patients/survivors will be asked to beta-test the cancer-specific app prototype for four weeks. The prototype will be developed in Aim 2 and informed by qualitative findings of Aim 1.
  Interventions: Device: Cancer-Specific Meditation App Prototype

INTERVENTIONS:
Other: Calm Meditation Smartphone App Feedback — Advisory committee members will be asked to use the current Calm meditation app platform for a full week and to keep an informal journal prior to participating in focus groups in which they will provide feedback about the app.
  Arms: Calm Meditation Smartphone App Feedback (Aim 1)
Other: Cancer-Specific Meditation App Prototype Design — Findings from Aim 1 will inform the development of a cancer-specific meditation app prototype to be tested in Aim 3.
  Arms: Cancer-Specific Meditation App Prototype Design (Aim 2)
Device: Cancer-Specific Meditation App Prototype — Recruited cancer patients/survivors will be asked to beta-test the cancer-specific app prototype for four weeks. The prototype will be developed in Aim 2 and informed by qualitative findings of Aim 1.
  Arms: Cancer-Specific Meditation App Prototype (Aim 3)

SUMMARY:
Using the IDEAS (Integrate, Design, Assess, and Share) framework, the investigators will conduct the following aims:

Specific Aim 1: Using two focus groups, the investigators will INTEGRATE formative work, the social cognitive theory, and perspectives from the experienced-user advisory committee (N=20) who will use the current Calm platform to identify design content and features for a standalone cancer-specific app prototype leveraging the commercial infrastructure of the Calm platform. The advisory committee will consist of both cancer patients/survivors (n=10; 5 of each) and health care providers (n=10).

Specific Aim 2: DESIGN a meditation app prototype tailored to cancer patients/survivors unique needs including content related to cancer-related experiences, emotions, symptoms, physical and psychological needs, cancer-specific symptom self monitoring, social support and sense of belonging within the app and through Facebook.

Specific Aim 3: ASSESS (i.e., beta-test) the prototype's form and function with cancer patients/survivors (N=30). The investigators will use Bowen's feasibility model to determine via surveys and interviews: (a) acceptability (satisfaction, perceived appropriateness, perceived positive/negative effects); (b) demand (use of the app, interest or intention to use); (c) practicality (how it makes them feel, ease of use); (d) adaptation (suggestions for modifications to improve performance for cancer patients/survivors); and (e) integration (how can the app be integrated into the cancer "system") Feasibility benchmarks: >80% of cancer patients/survivors will accept the prototype, demand the prototype for themselves and other cancer patients/survivors, and find it practical. Data from Aim 3 will guide refinement of the prototype to be tested in a fully powered RCT to establish long term engagement (Phase 2). This work will result in an evidence based, cancer-specific meditation app through a commercial platform that can be scaled and sold at discounted costs to clinic providers and directly to patients (SHARE; Phase 3).

DETAILED DESCRIPTION:
This STTR consists of three aims, each of which are conducted in successive order, with the end result being a cancer-specific meditation app prototype ready for efficacy testing (Phase 2) and direct marketing to the consumer (Phase 3).

Aim 1: Using the IDEAS framework, the investigators will INTEGRATE a) perspectives from an informed advisory committee (N=20) about the current Calm platform and b) strategies from the social cognitive theory to design a cancer-specific meditation app prototype. The meaning of the IDEAS stage INTEGRATE is to uncover deeper needs, values, and motivations, engaging key stakeholders (i.e., patients and providers) and use behavioral theory to inspire solutions that are more relevant and acceptable to the target population. Procedures: The advisory committee will consist of informed cancer patients, survivors (n=10; 5 of each) and healthcare providers (n=10; physicians, oncology nurses, cancer care coordinators, directors of integrative programs in cancer centers, and not-for-profit partners; See Support Letters). The advisory committee members are drawn from partnerships with Mays Cancer Center at UT Health San Antonio, MD Anderson, the Mayo Clinic in Scottsdale, AZ and Rochester, NY, University of Arizona, Wake Forest, Leukemia and Lymphoma Society, and the American Cancer Society. Both patients/survivors and providers are included on the advisory committee because providers play a key role in recommending mobile tools to patients to self-manage their symptoms, providers are often uninvolved stakeholders related to app design, and integrating apps into scalable interventions requires support of both patients/survivors and providers. The selection criteria prioritizes the cancer patient and survivor experience, but also includes members who see and hear the preferences, points of reluctance, stated and unstated barriers, and behavioral choices of those they serve in a variety of capacities (medical, ancillary, and direct provision of in-person meditation options).

The advisory committee will be asked to: (1) use the Calm app for at least 10 minutes a day for seven days to explore its content and features, (2) keep an informal journal of (a) time of day and time spent using Calm, (b) responses to app options and what motivated them to make certain choices, (c) their experiences during the guided meditations, and (d) ideas about life experiences of a cancer patient to include in prototype, (e) responses to prompts related to strategies from SCT, (e.g., in what ways might the content or features of the app support a sense of social modeling from other cancer patients or providers? How might goal setting and rewards be incorporated appropriately?) and (f) if not a cancer patient or survivor, to reflect upon the perspective of those they treat or serve, and (3) participate in a virtual focus group to provide informed, meaningful and specific input for the prototype. Focus groups have a long history in industry and marketing when the goal is to evaluate responses to products or ideas under development. Considering Coronavirus 2019, virtual focus groups will be conducted based on best-practice guidelines for internet-based qualitative research. One developer from Calm will listen to the focus groups for practical guidance and to meet target needs in the prototype design (Aim 2). The investigators will use Bowen's feasibility framework to explore specific domains of design (acceptability, demand, practicality, adaptation, and integration) (examples are open-ended experiential and cancer-referenced content explorations). The investigators believe this informed-user stage will strengthen the advisory committees' ability to direct the following design and assessment stages where they will be advisors not users. These informed-user focus groups will direct the DESIGN stage in Aim 2, by developing a list of the content and features, prioritized by numbers of mentions and importance emphasized. Milestone for Aim 1: Prioritize a list of 10-12 key content and feature issues to use in designing the prototype and promoting continued engagement.

Aim 2: Using the IDEAS framework, the investigators will DESIGN a cancer-specific meditation app prototype. IDEAS framework suggests prototyping leads to objectively stronger final products. The process includes understanding the most frequent requests, deciding on goals and non-goals, and writing out how users should interact with specific features. The investigators will use findings from Aim 1 to rapidly develop server-side Application Programming Interface (APIs) and an app for iOS. Themes and feedback from the feasibility focus groups (e.g., how to cultivate acceptance, demand, practicality, etc.) will be used to extend the current Calm design, APIs, and app so that the content, layout, and features in the app will address specific cancer-related long-term needs.

Design: The first step is to mock up user experience, user interface flows, and screens in the mobile app that fit with the values and user requirements from the focus groups. The investigators will mock and create wireframes of potential flow and solutions. The designs will be iterated based on feedback. Once the investigators have clear wireframes and specifications, they will create high-fidelity build mock ups.

API and mobile application development: The investigators will build out an interactive prototype by extending Calm's API. The API is a web interface that will help facilitate communication between the mobile application (front-end) and the software running on the server (back-end). It will allow the app to extend its functionalities by making use of other software subroutines running remotely on a server. The APIs will be REST-based and developed in JavaScript using a web framework known as Node.js with a Postgres database. The current Calm system is deployed using Kubernetes, provisioned with Terraform and hosted on Amazon Web Services. All API communication between the servers and clients is done through HTTPS (Hypertext Transfer Protocol Secure) for secure communication. The servers will handle the logic of what, where, when, and how information should be displayed. This will allow the front-end team to move more quickly, focus on user experience, user interface and beautiful animations rather than duplicating the complex business logic. The investigators can move very quickly to automatically change the way content is displayed on the server without user app updates. The API handles authentication, identity management, content, session history, subscriptions, AB test enrollment, assets, surveys and polls, onboarding flows, and scenes. The investigators also have admin endpoints that are deployed inside the virtual private cloud and are not publicly accessible. These routes power the internal tools, which support scene and program uploading, user management, admin activity logs and notes, and debugging. Thus, all aspects of the existing Calm app, from meditation tracks and content to the specific visual and selection paths, even to the inner structural workings of the app can be adapted with recommendations from Aim 1. After specifying the API changes, the investigators will change the API code and front-end app to speak to the API. This results in the prototype app specifically targeting cancer patients and survivors to be used in Aim 3. All data will be encrypted and the patient will use a password to access the app. Security and compliance standards will meet the requirements as a business associate of a healthcare provider, including HIPAA policies and procedures.

Aim 3: Using the IDEAS framework, the investigators will ASSESS (i.e., beta-test) the feasibility of the cancer-specific meditation app prototype with a sample of cancer patients/survivors (N=30). The investigators will recruit cancer patients/survivors with varying cancer types and stages, race/ethnicity, rural/urban geographic settings, and genders via social media. The investigators have 100 letters of support from cancer patients/survivors supporting the development of a cancer-specific Calm app. Studies suggest 5-10 participants are sufficient to establish feasibility and detect technical difficulties. The sample size is not to establish efficacy, but the multiple components of feasibility. The investigators have included a larger number to ensure a variety of cancer-related experiences. Beta-test participants will be asked to use the prototype for four weeks (free access) for at least 10 minutes per day, but will be encouraged to use it as much as they would like, mimicking how a new paying member would use the existing Calm app. Participation (meditations completed, time of day, length of time, components used) will be tracked (provided by Calm) over the four weeks. The 4-week period is not to establish efficacy but is an appropriate time to test feasibility. To determine acceptability, demand, and practicality, participants will be asked to complete weekly satisfaction questionnaires in addition to a final overall study satisfaction questionnaire immediately post-intervention using REDCap. Following the 4-week beta-test, and in addition to a satisfaction questionnaire the investigators will ask participants to volunteer for a semi-structured interview to determine, using Bowen's feasibility model, acceptability, demand, practicality, adaptation and integration to optimize potential for uptake, engagement and continued use at recommended levels (i.e., at least 10 min/day). Themes and findings from the interviews will be shared with the advisory committee and used to translate findings into app-relevant recommendations (i.e., further revisions if necessary) for efficacy testing (Phase 2). This approach is similar to methods used in other studies designing and developing mobile apps. Due to COVID-19, the investigators will conduct interviews virtually, based on best-practice guidelines for internet-based qualitative research.

ELIGIBILITY:
Interested cancer patients/survivors (Aim 3) will be asked to complete an eligibility survey via a REDCap survey link. Eligibility criteria is as follows:

Patients/survivors will be eligible if they are:

* at least 18 years of age
* able to read and understand English
* identify as a cancer patient (i.e., currently receiving treatment) or a survivor (i.e., prior patient no longer receiving treatment)
* willing to download the cancer-specific app prototype to their phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Aim 1: Feasibility: Acceptability as assessed with focus groups | Questions asked at one week of use of the current Calm platform
  Acceptability is defined as satisfaction, intent to continue to use, perceived appropriateness according to Bowen and colleagues feasibility criteria.
Feasibility: Demand as assessed with focus groups | Questions asked at one week of use of the current Calm platform
  Demand is defined as actual use, expressed interest or intention to use, perceived demand according to Bowen and colleagues feasibility criteria.
Aim 1: Feasibility: Practicality as assessed with focus groups | Questions asked at one week of use of the current Calm platform
  Practicality is defined as ability of participants to carry out intervention activities, efficiency/speed/quality of implementation according to Bowen and colleagues feasibility criteria.
Aim 1: Feasibility: Adaptation as assessed with focus groups | Questions asked at one week of use of the current Calm platform
  Adoption is defined as how to promote improvement according to Bowen and colleagues feasibility criteria.
Aim 1: Feasibility: Integration as assessed with focus groups | Questions asked at one week of use of the current Calm platform
  Integration is defined as Integration degree of execution, amount and type of resources needed to implement, factors affecting ease of implementation according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Acceptability as assessed with survey | Questions will be asked with a satisfaction survey after week 1
  Acceptability is defined as satisfaction, intent to continue to use, perceived appropriateness according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Acceptability as assessed with survey | Questions will be asked with a satisfaction survey after week 2
  Acceptability is defined as satisfaction, intent to continue to use, perceived appropriateness according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Acceptability as assessed with survey | Questions will be asked with a satisfaction survey after week 3
  Acceptability is defined as satisfaction, intent to continue to use, perceived appropriateness according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Acceptability as assessed with survey | Questions will be asked with a satisfaction survey after week 4
  Acceptability is defined as satisfaction, intent to continue to use, perceived appropriateness according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Acceptability as assessed with survey | Questions will be asked with a post-intervention (week 4) satisfaction survey
  Acceptability is defined as satisfaction, intent to continue to use, perceived appropriateness according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Acceptability as assessed with interview | Questions will be asked with a post-intervention (week 4) structured interview
  Acceptability is defined as satisfaction, intent to continue to use, perceived appropriateness according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Demand as assessed with survey | Questions will be asked with a satisfaction survey after week 1
  Demand is defined as actual use, expressed interest or intention to use, perceived demand according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Demand as assessed with survey | Questions will be asked with a satisfaction survey after week 2
  Demand is defined as actual use, expressed interest or intention to use, perceived demand according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Demand as assessed with survey | Questions will be asked with a satisfaction survey after week 3
  Demand is defined as actual use, expressed interest or intention to use, perceived demand according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Demand as assessed with survey | Questions will be asked with a satisfaction survey after week 4
  Demand is defined as actual use, expressed interest or intention to use, perceived demand according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Demand as assessed with survey | Questions will be asked with a post-intervention (week 4) survey
  Demand is defined as actual use, expressed interest or intention to use, perceived demand according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Demand as assessed with interview | Questions will be asked with a post-intervention (week 4) structured interview
  Demand is defined as actual use, expressed interest or intention to use, perceived demand according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Demand captured via Calm-provided data | Calm-provided data capturing meditation participation at post-intervention (week 4)
  Calm will track weekly minutes of meditation participation for each participant.
Aim 3: Feasibility: Practicality as assessed with survey | Questions will be asked with a satisfaction survey after week 1
  Practicality is defined as ability of participants to carry out intervention activities, efficiency/speed/quality of implementation according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Practicality as assessed with survey | Questions will be asked with a satisfaction survey after week 2
  Practicality is defined as ability of participants to carry out intervention activities, efficiency/speed/quality of implementation according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Practicality as assessed with survey | Questions will be asked with a satisfaction survey after week 3
  Practicality is defined as ability of participants to carry out intervention activities, efficiency/speed/quality of implementation according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Practicality as assessed with survey | Questions will be asked with a satisfaction survey after week 4
  Practicality is defined as ability of participants to carry out intervention activities, efficiency/speed/quality of implementation according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Practicality as assessed with survey | Questions will be asked with a post-intervention (week 4) survey
  Practicality is defined as ability of participants to carry out intervention activities, efficiency/speed/quality of implementation according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Practicality as assessed with interview | Questions will be asked with a post-intervention (week 4) structured interview
  Practicality is defined as ability of participants to carry out intervention activities, efficiency/speed/quality of implementation according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Adaptation as assessed with survey | Questions will be asked with a weekly satisfaction survey (week 1 to week 4)
  Adoption is defined as how to promote improvement according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Adaptation as assessed with survey | Questions will be asked with a satisfaction survey after week 1
  Adoption is defined as how to promote improvement according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Adaptation as assessed with survey | Questions will be asked with a satisfaction survey after week 2
  Adoption is defined as how to promote improvement according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Adaptation as assessed with survey | Questions will be asked with a satisfaction survey after week 3
  Adoption is defined as how to promote improvement according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Adaptation as assessed with survey | Questions will be asked with a satisfaction survey after week 4
  Adoption is defined as how to promote improvement according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Adaptation as assessed with interview | Questions will be asked with a post-intervention (week 4) structured interview
  Adoption is defined as how to promote improvement according to Bowen and colleagues feasibility criteria.
Aim 3: Feasibility: Integration as assessed with survey | Questions will be asked with a post-intervention (week 4) survey
  Integration is defined as Integration degree of execution, amount and type of resources needed to implement, factors affecting ease of implementation according to Bowen and colleagues feasibility criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Calm, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huberty J, Bhuiyan N, Puzia M, Joeman L, Larkey L, Mesa R. Meditation Mobile App Developed for Patients With and Survivors of Cancer: Feasibility Randomized Controlled Trial. JMIR Cancer. 2022 Nov 23;8(4):e39228. doi: 10.2196/39228. PMID 36416880